CLINICAL TRIAL: NCT00145106
Title: Regimen of Tazorac .1% Gel & Minocycline Cap in Tx of Individuals w/Acne Vulgaris: Effects of Maintenance Therapy on Duration of Improvement of Tazorac .1% Gel Used in Conjunction w/Placebo Cap Compared w/Minocycline Cap Used in Conjunction w/Either Tazorac .1% Gel or Vehicle Gel
Brief Title: Comparison of Tazarotene and Minocycline Therapies for Maintenance of Facial Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KGL, Inc. (Other)
Collaborators: Milton S. Hershey Medical Center (Other); State University of New York - Downstate Medical Center (Other); Jefferson Medical College of Thomas Jefferson University (Other); NYU Langone Health (Other); Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T214
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-09

CONDITIONS: Acne Vulgaris
Keywords: acne, tazarotene, minocycline, maintenance, retinoid, efficacy, combination
MeSH Terms: conditions — Acne Vulgaris; cyclopia sequence | interventions — tazarotene; Gels; Minocycline; Capsules

INTERVENTIONS:
Drug: Tazarotene 0.1% gel + placebo capsule, Oral minocycline (100 mg capsule) + vehicle gel, Tazarotene 0.1% gel + oral minocycline (100 mg capsule)

SUMMARY:
The purpose of the study is to compare the efficacy of three maintenance regimens (topical tazarotene, oral minocycline, or both) in sustaining improvement in acne.

DETAILED DESCRIPTION:
For many years antibiotic therapy has been the backbone of therapy for inflammatory acne. However, topical retinoids also offer efficacy against inflammatory acne and the combination of a topical retinoid and an antibiotic can result in faster and more complete clearing of inflammatory lesions than either drug alone.

The reduced sensitivity of Propionibacterium acnes to antibiotics is a growing problem. Resistance is a major issue not only because it can result in treatment failure but also because of concerns that it may potentially be transferred to other bacteria that anti-acne antibiotics are used used against. One of the most important factors predisposing to the development of resistant strains of propionibacterium acnes is the prolonged use of antibiotics. Therefore, in order to help minimize the development for such resistance, it is evident that maintenance strategies for acne should aim to minimize the long-term use of antibiotics.

Topical retinoids are a rational choice for maintenance therapy due to their activity on microcomedones (the precursor for all acne lesions). Nevertheless, there is a paucity of data evaluating this use in a maintenance setting. The aim of this study was to determine whether patients with moderate to severe inflammatory acne who have achieved a good level of clearance (eg>/= 75%) can maintain the improvement in their acne using maintenance therapy. THe study compared the efficacy of three maintenance therapies (topical tazarotene, oral minocycline, and topical tazarotene plus oral minocycline) in sustaining the clinical improvement attained after initial topical tazarotene plus oral minocycline therapy.

ELIGIBILITY:
Inclusion Criteria:

Moderate facial acne vulgaris 25-60 facial inflammatory acne lesions 10-100 facial comedos No more than 2 facial nodular cystic lesions (no more than 5 mm in diameter) For females of child bearing potential, a regular menstrual cycle Negative urine pregnancy test

Exclusion Criteria:

Uncontrolled systemic disease Acne vulgaris known to be resistant to antibiotics For females: pregnancy, breastfeeding, or planning pregnancy Use of estrogens or birth control pills for 12 weeks or less Any skin disease that may interfere with diagnosis or evaluation of acne vulgaris Known hypersensivity to any components in Tazarac gel or to any tetracyclines Use of any systemic retinoids in past 2 years Use of any systemic antibiotics, or participation in another drug or investigational study, in past 30 days Use of topical anti-acne medication in past 14 days

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189
Dates: Start 2002-03; Study Completion 2002-08

PRIMARY OUTCOMES:
Global improvement from baseline at week 24

SECONDARY OUTCOMES:
Lesion counts at weeks 16, 20 and 24

CONTACTS AND LOCATIONS:
Overall Officials: James Leyden, MD, Principal Investigator — KGL, Inc.
Locations (1):
- KGL, Inc, Broomall, Pennsylvania, United States